CLINICAL TRIAL: NCT00608725
Title: Pathophysiology of Orthostatic Intolerance
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Satish R. Raj (Other)
Responsible Party: Sponsor-Investigator, Satish R. Raj, Assistant Professor of Medicine & Pharmacology, Vanderbilt University Medical Center
Organization: Vanderbilt University Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 8398
Record Dates: First submitted 2008-01-22; First posted 2008-02-06 (Estimated); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Tachycardia; Postural Orthostatic Tachycardia Syndrome
Keywords: heart rate; blood pressure; blood volume; sympathetic nervous system; orthostatic tachycardia; orthostatic intolerance; POTS
MeSH Terms: conditions — Tachycardia; Postural Orthostatic Tachycardia Syndrome; Orthostatic Intolerance | interventions — Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients (Other): Patients with orthostatic intolerance
  Interventions: Radiation: DAXOR; Procedure: QSweat; Drug: Intrinsic Heart Rate
- Healthy Control Subjects (Other): Healthy subjects to determine "normal" response
  Interventions: Radiation: DAXOR; Procedure: QSweat; Drug: Intrinsic Heart Rate

INTERVENTIONS:
Radiation: DAXOR — 131-I-Human Serum Albumin Blood Volume Assessment Kit
  Other Names: Volumex
Procedure: QSweat — Quantitative Sweat Testing
  Other Names: QSART; Quantitative Axonal Sudomotor Reflex Testing
Drug: Intrinsic Heart Rate — Atropine 0.04 mg/kg IV in divided doses Propranolol 0.2 mg/kg IV in divided doses
  Other Names: Inderal; IHR

SUMMARY:
The purpose of this study is to describe the mechanism of orthostatic intolerance, relying on cardiovascular physiological studies. The syndrome is of undetermined etiology, but the syndrome causes impairment of a number of young adults, females more than males, with symptoms of tachycardia, fatigue, lightheadedness, palpitations, blurred vision, chest discomfort, difficulty concentrating, and dizziness with the upright posture. It is believed that many different pathophysiological processes can give rise to this disorder.

DETAILED DESCRIPTION:
The purpose of this study is to describe the mechanism of orthostatic intolerance, relying on cardiovascular physiological studies. The syndrome is of undetermined etiology, but the syndrome causes impairment of a number of young adults, females more than males, with symptoms of tachycardia, fatigue, lightheadedness, palpitations, blurred vision, chest discomfort, difficulty concentrating, and dizziness with the upright posture. It is believed that many different pathophysiological processes can give rise to this disorder.

This is not a clinical trial in the classical sense, but an omnibus protocol to allow for disntinct and personalized pathophysiological testing.

ELIGIBILITY:
Inclusion Criteria:

* Orthostatic intolerance

Exclusion Criteria:

* Inability or unwillingness to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 1996-12; Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Physiological abnormalities in orthostatic intolerance | 1 day
  varied metrics used here

SECONDARY OUTCOMES:
blood volume | 1 day
  Blood volume as measured by DAXOR technique
intrinsic heart rate | 1 hour
  Heart rate after IV propranolol and IV atropine
quantitative sweat testing | 2 hours
  sweat volumes after a QSweat test
residual sympathetic function after pharmacological autonomic blockade | 3 hours
  changes in BP after trimethaphan infusions
norepinephrine spillover | 3 hours
  tritiated norepunephrine spillover data

CONTACTS AND LOCATIONS:
Overall Officials: David Robertson, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Mustafa HI, Garland EM, Biaggioni I, Black BK, Dupont WD, Robertson D, Raj SR. Abnormalities of angiotensin regulation in postural tachycardia syndrome. Heart Rhythm. 2011 Mar;8(3):422-8. doi: 10.1016/j.hrthm.2010.11.009. Epub 2011 Jan 22. PMID 21266211
- See also: Website of the Vanderbilt Autonomic Dysfunction Center — https://www.vumc.org/autonomic-dysfunction-center/vanderbilt-autonomic-dysfunction